CLINICAL TRIAL: NCT03933137
Title: Correlation Between P-POSSUM Score and Length of Stay in Kidney Transplant Recipients
Brief Title: P-POSSUM Score and Length of Stay
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, MD, PhD, Anesthesiologist Consultant, Indonesia University
Other Study IDs: IndonesiaUAnes034
Record Dates: First submitted 2019-04-24; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Length of Stay
Keywords: mortality; morbidity; length of stay; kidney; transplant
MeSH Terms: interventions — Morbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Not prolonged length of stay: Living donor patients who had ≤ 6 days length of stay after laparoscopic nephrectomy procedure
  Interventions: Other: Portsmouth Physiological and Operative Severity Score for the Enumeration of Mortality and Morbidity (P-POSSUM) score
- Prolonged length of stay: Living donor patients who had > 6 days length of stay after laparoscopic nephrectomy procedure
  Interventions: Other: Portsmouth Physiological and Operative Severity Score for the Enumeration of Mortality and Morbidity (P-POSSUM) score

INTERVENTIONS:
Other: Portsmouth Physiological and Operative Severity Score for the Enumeration of Mortality and Morbidity (P-POSSUM) score — P-POSSUM score's variables are divided into physiological parameters (age, cardiac, respiratory, ECG, systolic blood pressure, pulse rate, haemoglobin, leukocyte count, urea, sodium plasma, potassium plasma, and GCS) and operative parameters (operation type, number of procedures, operative blood loss, peritoneal contamination, malignancy status, CEPOD).

SUMMARY:
P-POSSUM score had a predictive power of >80% to predict the length of stay of kidney transplant recipients

ELIGIBILITY:
Inclusion Criteria:

* Subjects are medical record of recipients who underwent kidney transplant

Exclusion Criteria:

* Medical record was incomplete
* Patients who died during surgery or before the patient was discharged.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical record of recipients who undewernt kidney transplant during a period between January 2015 and December 2017
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Correlation between each variable of P-POSSUM and length of stay | 1 day before surgery until discharged from hospital, up to 30 days
  Correlation between 18 variables (12 variables as physical parameters and 6 variables as operative parameters) and length of stay
P-POSSUM score Discrimination | 1 day before surgery until discharged from hospital, up to 30 days
  P-POSSUM score ability to discriminate length of stay based on variable scores: physical parameters and operative parameters
P-POSSUM score Calibration | 1 day before surgery until discharged from hospital, up to 30 days
  P-POSSUM score cutoff to predict length of stay based on variable scores: physical parameters and operative parameters

SECONDARY OUTCOMES:
Patient's length of stay post kidney transplantation | From post surgery until discharged from hospital, up to 30 days
  Patient's length of stay post kidney transplantation
P-POSSUM score (physical parameters): Age | 1 day before surgery
  The score for Age variable cut-off:
  1. point for <61 years
  2. point for 61-71 years
  4 point >71 years
P-POSSUM score (physical parameters): Heart disease | 1 day before surgery
  The score for heart disease variable cut-off:
  1. point for no heart failure
  2. point for diuretic, digoxin or angina/hypertension medicine usage
  4 point for peripheral edema, warfarin, or borderline cardiomegaly on chest X-ray (CXR)
P-POSSUM score (physical parameters): Lung disease | 1 day before surgery
  The score for lung disease variable cut-off:
  1. point for no dyspnea
  2. points for exertional dyspnea or mild COPD on CXR
  4 points for limiting dyspnea or moderate COPD on CXR 8 points for dyspnea at rest or fibrosis/consolidation on CXR
P-POSSUM score (physical parameters): ECG abnormality | 1 day before surgery
  The score for ECG abnormality variable cut-off:
  1 point for normal ECG 4 points for atrial fibrillation (HR 60-90 8 points for 5 ectopic beats/min, Q waves or ST/T wave change
P-POSSUM score (physical parameters): Systolic blood pressure | 1 day before surgery
  The score for systolic blood pressure variable cut-off:
  1. point for 110 - 130 mmHg
  2. points for 100-109 mmHg or 131-170 mmHg
  4 points for > 170 mmHg or 90-99 mmHg 8 points for < 90 mmHg
P-POSSUM score (physical parameters): Pulse rate | 1 day before surgery
  The score for pulse rate variable cut-off:
  1. point for 50-80 beats per minute (bpm)
  2. points for 40-59 bpm or 81-100 bpm
  4 points for 101-120 bpm 8 points for > 121 bpm or < 40 bpm
P-POSSUM score (physical parameters): Hemoglobin | 1 day before surgery
  The score for hemoglobin variable cut-off:
  1. point for 13-16 g/dL
  2. points for 11.5-12.9 or 16.1-17 d/dL
  4 points for 10-11.4 or 17.1-18 g/dL 8 points for <10 or >18 g/dL
P-POSSUM score (physical parameters): Leukocyte count | 1 day before surgery
  The score for leukocyte count variable cut-off:
  1. point for 4.000-10.000/mm3
  2. points for 10.100-20.000 atau 3.100-4.000/mm3
  4 points for >20.000 atau <3.000/mm3
P-POSSUM score (physical parameters): Plasma potassium concentration | 1 day before surgery
  The score for plasma potassium concentration variable cut-off:
  1. point for 3.5-5 mmol/L
  2. points for 3.2-3.4 or 5.1-5.3 mmol/L
  4 points for 2.9-3.1 or 5.4-5.9 mmol/L 8 points for <2.9 or >5.9 mmol/L
P-POSSUM score (physical parameters): Plasma sodium concentration | 1 day before surgery
  The score for plasma sodium concentration variable cut-off:
  1. point for >135 mmol/L
  2. points for 131-135 mmol/L
  4 points for 126-130 mmol/L 8 points for <126 mmol/L
P-POSSUM score (operative parameters): Number of procedures | 1 day before surgery
  The score for number of procedures variable cut-off:
  1 point for one 4 points for two 8 points for more than two
P-POSSUM score (operative parameters): Intraoperative blood loss | Intraoperative
  The score for intraoperative blood loss variable cut-off:
  1. point for <100 mL
  2. points for 101-500 mL
  4 points for 501-999 mL 8 points for > 999 mL
P-POSSUM score (operative parameters): Peritoneal contamination/soiling | Intraoperative
  The score for peritoneal contamination/soiling variable cut-off:
  1. point for none
  2. points for minor (serous fluid)
  4 points for local pus 8 points for free bowel content, pus or blood
P-POSSUM score (operative parameters): Presence of malignancy | 1 day before surgery
  The score for presence of malignancy variable cut-off:
  1. point for none
  2. points for primary only
  4 points for nodal metastases 8 points for distant metastases
P-POSSUM score (operative parameters): Mode of surgery | 1 day before surgery
  The score for mode of surgery variable cut-off:
  1 point for elective 4 points for emergency resuscitation of > 2 hours possible operation < 24 hours after admission 8 points for emergency (immediate surgery < 2 hours needed)

CONTACTS AND LOCATIONS:
Overall Officials: Dita Aditianingsih, M.D, PhD, Study Chair — Department of Anesteshiology and Intensive Care, Cipto Mangunkusumo Hospital, Universitas Indonesia
Locations (1):
- Rumah Sakit Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Reyna-Sepulveda F, Ponce-Escobedo A, Guevara-Charles A, Escobedo-Villarreal M, Perez-Rodriguez E, Munoz-Maldonado G, Hernandez-Guedea M. Outcomes and Surgical Complications in Kidney Transplantation. Int J Organ Transplant Med. 2017;8(2):78-84. Epub 2017 May 1. PMID 28828167
- [Background] Howes TE, Cook TM, Corrigan LJ, Dalton SJ, Richards SK, Peden CJ. Postoperative morbidity survey, mortality and length of stay following emergency laparotomy. Anaesthesia. 2015 Sep;70(9):1020-7. doi: 10.1111/anae.12991. Epub 2015 Apr 15. PMID 25872411
- [Background] McAdams-DeMarco MA, King EA, Luo X, Haugen C, DiBrito S, Shaffer A, Kucirka LM, Desai NM, Dagher NN, Lonze BE, Montgomery RA, Walston J, Segev DL. Frailty, Length of Stay, and Mortality in Kidney Transplant Recipients: A National Registry and Prospective Cohort Study. Ann Surg. 2017 Dec;266(6):1084-1090. doi: 10.1097/SLA.0000000000002025. PMID 27655240
- [Background] Khambalia HA, Moinuddin Z, Summers AM, Tavakoli A, Pararajasingam R, Campbell T, Dhanda R, Forgacs B, Augustine T, van Dellen D. A prospective cohort study of risk prediction in simultaneous pancreas and kidney transplantation. Ann R Coll Surg Engl. 2015 Sep;97(6):445-50. doi: 10.1308/rcsann.2015.0001. Epub 2015 Aug 14. PMID 26274754
- [Background] Grocott MP, Levett DZ, Matejowsky C, Emberton M, Mythen MG. ASA scores in the preoperative patient: feedback to clinicians can improve data quality. J Eval Clin Pract. 2007 Apr;13(2):318-9. doi: 10.1111/j.1365-2753.2006.00736.x. No abstract available. PMID 17378882
- [Background] Chen T, Wang H, Wang H, Song Y, Li X, Wang J. POSSUM and P-POSSUM as predictors of postoperative morbidity and mortality in patients undergoing hepato-biliary-pancreatic surgery: a meta-analysis. Ann Surg Oncol. 2013 Aug;20(8):2501-10. doi: 10.1245/s10434-013-2893-x. Epub 2013 Feb 23. PMID 23435569
- [Background] Moonesinghe SR, Mythen MG, Das P, Rowan KM, Grocott MP. Risk stratification tools for predicting morbidity and mortality in adult patients undergoing major surgery: qualitative systematic review. Anesthesiology. 2013 Oct;119(4):959-81. doi: 10.1097/ALN.0b013e3182a4e94d. PMID 24195875
- [Background] Baron DM, Hochrieser H, Posch M, Metnitz B, Rhodes A, Moreno RP, Pearse RM, Metnitz P; European Surgical Outcomes Study (EuSOS) group for Trials Groups of European Society of Intensive Care Medicine; European Society of Anaesthesiology. Preoperative anaemia is associated with poor clinical outcome in non-cardiac surgery patients. Br J Anaesth. 2014 Sep;113(3):416-23. doi: 10.1093/bja/aeu098. Epub 2014 May 14. PMID 24829444
- [Background] Li S, Zhou K, Lai Y, Shen C, Wu Y, Che G. Estimated intraoperative blood loss correlates with postoperative cardiopulmonary complications and length of stay in patients undergoing video-assisted thoracoscopic lung cancer lobectomy: a retrospective cohort study. BMC Surg. 2018 May 23;18(1):29. doi: 10.1186/s12893-018-0360-0. PMID 29792183
- [Background] Amer MS, Hamza SA, Wahba HMF, Barakat DB. Effects of Anemia on The Outcome in Elderly Admitted to The ICU. Indian J Med Res Pharm Sci. 2016;3(April):27-32.